CLINICAL TRIAL: NCT00259857
Title: A Randomized, Double-Blind, Placebo-Controlled, Prospective, Cross-Over Phase II Clinical Trial to Determine the Safety and Efficacy of Alendronate (Fosamax) in Juvenile Osteoporosis (IND#60,017)
Brief Title: Safety and Efficacy of Alendronate (Fosamax) in Children With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Deborah A Bowlby, MD, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01FD001847-05 (FDA); FDR00184705-83045-05 (Other: Medical University of South Carolina)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-12

CONDITIONS: Osteoporosis
Keywords: Fracture; Bone Mineral Density; DXA
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Alendronate; Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Alendronate, Calcium, Vitamin D (Experimental): Crossover study. Year-1, 10 participants will take study medication, calcium and vitamin D supplements and other 10 participants will take placebo, calcium and vitamin D supplements. Year-2, they will crossover to the second arm of the study. Those who took study medication and supplements in year-1, will take placebo and supplements in the year-2, and those 10 participants who took placebo and supplements in the year-1, will take study medications and supplements in the year-2.
  Interventions: Drug: Alendronate
- 2 Placebo, Calcium and Vitamin D (Placebo Comparator): Year-1, 10 participants will take Alendronate (study medication)and calcium and vitamin D supplement). Another 10 participants will take placebo, calcium and vitamin D. In year-2 they will crossover. Those who took alendronate in the first year, will take Placebo, calcium and vitamin D for 12 months and those who took Placebo in the first year, will take Alendronate, calcium and vitamin D in the second year (12 months).
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Group-1/Year-1:Alendronate, pill, 35mg or 70mg, weekly; calcium, pill, 500mg or 1000mg daily; vitamin D, liquid, 800IU, daily, depending upon the body weight, for 12 months. Group-1/Year-2:Placebo, pill, 35mg or 70mg, weekly; calcium, pill, 500mg or 1000mg daily; vitamin D, liquid, 800IU, daily, depending upon the body weight for 12 months. Group-2/Year-1:Placebo, pill, 35mg or 70mg, weekly; calcium, pill, 500mg or 1000mg daily; vitamin D, liquid, 800IU, daily, depending upon the body weight for 12 months. Group-2/Year-2: Alendronate, pill, 35mg or 70mg, weekly; calcium, pill, 500mg or 1000mg daily; vitamin D, liquid, 800IU, daily, depending upon the body weight for 12 months.
  Other Names: Fosamax; TUMS or Viactive; Drisdol or Calciferol

SUMMARY:
We have previously evaluated the safety and efficacy of Alendronate in 10 patients with juvenile osteoporosis during a 12-month clinical trial. We have documented that Alendronate improved BMD of the spine and hip without any major side effects. There were no additional fractures during therapy. The present study is designed to further evaluate the safety and efficacy of Alendronate in 20 children with juvenile osteoporosis using a double-blind, randomized, placebo-controlled, cross-over protocol.

DETAILED DESCRIPTION:
Osteoporosis is an uncommon disease in children and early adolescents. Patients have a low bone mineral density, develop fractures with minimal or no trauma, and frequently have a negative family history. The disease results from either diminished bone formation or increased bone removal (resorption). No specific drug therapy has been recommended for juvenile osteoporosis. Alendronate (Fosamax) is effective in inhibiting bone resorption, increasing BMD and reducing fractures in adults with postmenopausal osteoporosis, but have not become established therapies in children. In the present study, we plan to evaluate the safety and efficacy of Alendronate in 20 patients with juvenile osteoporosis in a two-year period. This is a randomized, double-blind, placebo-controlled protocol. In the year-1, 10 patients will be assigned to receive Alendronate and 10 patients placebo. In the year-2, patients will be crossed over to the second arm of the study. Those who received Alendronate in the year-1, will receive placebo in the second year and vice verse. The patients will have 5 visits, the initial screening visit followed by 4 post therapy visits in a six-month interval. Measurements include DXA bone density scan of spine and hip, urinalysis and blood work.

ELIGIBILITY:
Eligibility Criteria:

* 5-15 yrs of age
* Weighing 20 kg and more
* History of multiple fractures
* Tanner stage II or less
* Osteoporosis by DXA.

Inclusion Criteria:

* Male and female children with a history of one or more atraumatic fractures, or evidence of one or more compression fractures on radiographs of the spine (reduction of >20 percent).
* Bone Mineral Density (BMD) determined by DXA sacn to confirm osteoporosis at a Z score greater than 2 SD (standard deviations) below the normal mean for age (Z score < -2 SD).
* Parental consent (and patient assent after age 12 years) to participate in the study.
* Sexual development at: Tanner stage II or less (Prepubertal stage).
* Weight = 20 kg and more.

Exclusion Criteria:

* History of severe gastritis or reflux.
* Abnormalities of the esophagus that delay emptying, such as strictures or achalasia
* Marked kyphoscoliosis or the inability to sit or stand for at least 30 minutes
* Hypersensitivity to bisphosphonates
* Uncorrected hypocalcemia
* History of gastric or duodenal ulcers
* Renal dysfunction as indicated by serum Cr >1.5 mg/dl.
* Liver dysfunction as indicated by serum SGPT > 2 times the upper limit for age or serum total bilirubin > 2.0 mg/dl.
* Diagnosis of osteogenesis imperfecta, a family history of osteogenesis imperfecta, blue sclerae or deafness.
* Diagnosis of active rickets or osteomalacia or serum bone alkaline phosphatase 2 times greater than normal for age.
* Pregnancy
* Anorexia Nervosa

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2003-10; Primary Completion 2008-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Bowlby, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Key LL Jr, Ries W, Madyastha P, Reed F. Juvenile osteoporosis: recognizing the risk. J Pediatr Endocrinol Metab. 2003 May;16 Suppl 3:683-6. PMID 12795371
- See also: Medical University of South Carolina, Children's Hospital — http://www.musckids.com/research/fosamax_trial.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period:O5/27/2004 to 02/01/2006. Types of location:outpatient clinic, Clinical and Translational Research Center (CTRC), Medical University of South Carolina, Charleston, South Carolina.
Groups:
- Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D: Group-1/Year-1, 11 participants will take Alendronate,(study medication) and calcium, and vitamin D (supplements) and in Year-2 they will crossover to placebo, calcium and vitamin D supplements.
- Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D: Group-2/Year-1, 11 participants will take Placebo,and calcium, and vitamin D (supplements) and in Year-2 they will crossover to Alendronate (study medication), calcium and vitamin D (supplements).
Period: 12 Months Treatment
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2
Not completed — Gr-1, lost followup; Gr-2, not compliant | 1 | 2
Period: 24 Months Treatment
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Started | 10 | 9
Completed | 10 | 6
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.17 (2.8) | 9.47 (2.3) | 9.32 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Bone Mineral Density (BMD) of Spine After Therapy
Description: Participants were screened for BMD of lumbar spine using DXA scan at visit 12 months after alendronate or placebo treatment.
Time Frame: 12 months therapy
Population: Analysis was done per protocol and intention to treat.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 10 | 9
participants | 10 | 9

2. Secondary Outcome: Number of Participants With Improvement in Bone Mineral Density (BMD) of Hip After Therapy
Time Frame: 12 months of therapy
Population: Analysis was done per protocol and intention to treat.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 10 | 9
participants | 10 | 9

3. Primary Outcome: Number of Participants With Improvement in Bone Mineral Density (BMD) of Spine After Therapy
Description: BMD of lumbar spine was measured using DXA scan at visit 24 months (Year-2)after alendronate or placebo treatment.
Time Frame: 24 months therapy
Population: Analysis was done per protocol and intention to treat.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 10 | 6
participants | 10 | 6

4. Secondary Outcome: Number of Participants With Improvement in BMD of Hip
Description: Analysis was done per protocol and intention to treat.
Time Frame: 24 months of therapy
Population: Analysis was done per protocol and intention to treat.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 10 | 6
participants | 10 | 6

5. Secondary Outcome: Participants With Atraumatic Fractures
Description: Number of Participants with Atraumatic fractures before therapy.
Time Frame: 0 months
Population: Number of participants with fractures before therapy.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 11 | 11
participants | 11 | 11

6. Secondary Outcome: Participants With Atraumatic Fractures
Description: Number of participants with fractures at the completion of therapy.
Time Frame: 24 months
Population: Number of participants with fractures at study completion.
Measure: Number; unit: participants
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Number analyzed (Participants) | 10 | 6
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: two years
Description: To make monthly phone calls to assess any side effects or adverse events.
Arm/Group | Gr-1:Yr-1/Yr-2: Alendronate/Pbo, Calcium, Vitamin D | Gr-2:Yr-1/Yr-2: Pbo/Alendronate, Calcium and Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement with Merck: to submit a copy of any proposed abstract, manuscript and/or press release to Merck for review and comment at least 30 days prior to submission for publication or presentation.